CLINICAL TRIAL: NCT05031052
Title: Normothermic Machine Perfusion (NMP) Compared to Static Cold Storage (SCS) in Donation After Brain Death (DBD) Kidney Transplantation; a Prospective Multicenter Randomized Controlled Trial (NMP-DBD)
Brief Title: Normothermic Machine Perfusion (NMP) Versus Static Cold Storage (SCS) in Human Kidney Transplantation
Acronym: NMP-DBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Georg Lurje, MD, Consultant HPB- and Transplant Surgeon, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA4/172/21
Record Dates: First submitted 2021-08-23; First posted 2021-09-01 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Kidney Transplant; Complications; Kidney Failure; Graft Dysfunction
Keywords: ex-vivo machine perfusion; normothermic machine perfusion; kidney transplantation; extended criteria donation; donation after brain death; NMP
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normothermic machine perfusion (NMP) (Experimental): End-ischemic NMP will be performed immediately after arrival of the allocated and static cold stored ECD kidney graft. The study protocol aims a duration of 4 hours. Machine perfusion will be performed with a combination of patient's blood group matched packed red blood cells (RBC) and a special manufactured solution with the currently only certified device in Europe (XVIVO - KidneyAssist®). After 4 hours of perfusion and viability assessment, the kidney allograft will be disconnected from the device immediately prior to transplantation and flushed with three litres of Custodiol HTK solution via the renal artery. Then transplantation will be performed in typical method.
  Interventions: Device: End-ischemic normothermic oxygenated machine perfusion
- Statical cold storage (SCS) (Active Comparator): Conventional method kidney transplantation of statical cold stored and transported ECD kidney allograft. The allocated kidney allograft will be flushed with Custodiol HTK solution during back table preparation with the aim of immediate implantation into recipient.
  Interventions: Procedure: Static cold storage

INTERVENTIONS:
Device: End-ischemic normothermic oxygenated machine perfusion — Application of end-ischemic normothermic oxygenated machine perfusion at physiological temperatures for 4 hours.
  Other Names: NMP
  Arms: Normothermic machine perfusion (NMP)
Procedure: Static cold storage — Immediate implantation of kidney allograft after conventional and static preservation on ice
  Other Names: SCS
  Arms: Statical cold storage (SCS)

SUMMARY:
Due to organ shortage in kidney transplantation (KT) several strategies have been implemented in an attempt to increase donor pool utilization, including transplantation of extended criteria donor (ECD) allografts. While the transplantation of ECD organs saves patients from waiting-list dropout, these pre-damaged organs exhibit an increased susceptibility to further injury during organ storage and transplantation. Static cold storage (SCS) involves the transportation of procured donor kidneys on ice and has remained the gold standard for organ preservation for decades. SCS relies on hypothermia to reduce cellular metabolism and oxygen demand while achieving a prolonged preservation time of organs. Upon reperfusion, the reintroduction of oxygen to the ischemic kidney leads to a respiratory burst with massive production of mitochondrial reactive oxygen species and subsequent sterile inflammation of the entire organ. This ischemia-reperfusion injury (IRI) is a central predictor of graft and patient survival. Current clinical preservation strategies are unable to meet the challenges of ECD allograft transplantation and there is a great demand to optimize preservation techniques for such high risk ECD allografts.

Currently, two main paradigms prevail in the clinical approach to kidney allograft machine perfusion (MP) in regard to optimized preservation techniques: while end-ischemic hypothermic (HMP) and hypothermic oxygenated MP (HOPE) may be seen as dynamic alternatives of the traditional organ preservation based on hypothermia-induced deceleration of metabolism could not proof a beneficial effect on delayed graft function or primary graft failure, the impact of normothermic perfusion (NMP) on ECD kidney allografts is still missing. NMP aims at re-equilibration of cellular metabolism by preserving the organ at physiological temperatures whilst ensuring sufficient oxygen and nutrient supply. The present trial was therefore designed to provide first level-II evidence for NMP in human KT after donation after brain death (DBD). In total, 194 human kidney grafts will be randomized to either 4 hours of NMP directly before implantation (intervention group; n = 97) or to SCS (control group; n = 97) prior to transplantation. The primary endpoint will be kidney function after 6 months (6-months eGFR). Secondary endpoints include kidney function after 3 and 12 months, incidence of delayed graft function (DGF), primary non-function (PNF) and surgical complications assessed by the comprehensive complication index (CCI).

DETAILED DESCRIPTION:
The first human kidney transplantation (KT) was performed by Murray et al. in 1954 and has evolved as the standard treatment for kidney failure (previously referred to as end-stage renal disease (ESRD). In 2020, approximately 7067 patients were listed for KT in Germany, however only 1342 transplantations could be performed due to organ shortage. The number of patients on the waiting list substantially exceeds the number of donors. Around 390 patients died while waiting for a suitable organ on the waiting list, and another 492 patients dropped out due to morbidity and advancing disease. For increasing donor pool utilization several strategies have been aimed, including living donation, old-for-old KT and transplantation of extended criteria donor (ECD) allografts. While, ECD allografts are associated with a higher incidence of graft related complications and impaired postoperative outcome, novel preservation techniques such as ex-vivo machine perfusion (MP) of the donor allograft have been developed aiming at optimizing the function of marginal organs after transplantation.

The common practice of static cold storage (SCS) organ preservation has changed little since the initial introduction of the original University of Wisconsin (UW) organ preservation solution in the late 1980s. Static organ preservation relies on hypothermia to decelerate metabolism and reduce oxygen demand to prolong ischemia tolerance and avoid rapid functional graft impairment, thereby delaying graft damage. While a significant amount of anaerobic metabolism continues at a low rate, the metabolism of the allograft does not cease completely during SCS. In addition, the lack of blood flow-derived shear stress causes a disruption of endogenous nitric-oxide (NO) production and a functional impairment of endothelial cells. Upon reperfusion, the reintroduction of oxygen-rich blood to the ischemic allograft leads to a respiratory-burst with massive reactive oxygen species (ROS) production, mitochondrial oxidative stress and a sterile inflammatory reaction that is pivotal to kidney injury. This cascade of ischemia-reperfusion injury (IRI) ultimately leads to an impaired outcome, especially in the ECD-KT setting. While high-quality grafts are usually less prone to IRI, ECD allografts exhibit an impaired microcirculation and an increased susceptibility to inflammatory and oxidative stress and, as such, poorly tolerate extended periods of cold storage.

In recent years, MP has been recognized as a promising strategy in the context of ECD kidney transplantation. While SCS only prolongs storage time and limits the damage sustained during the period of cold ischemia, MP can reverse some of these effects.

Hypothermic (HMP) and hypothermic oxygenated MP (HOPE) may be seen as dynamic cold organ preservation based on hypothermia-induced deceleration of metabolism, which aims to combine the positive effects of hypothermia observed in classical cold storage with the positive effects of dynamic preservation. In contrast normothermic perfusion (NMP) mimics physiological circumstances and provides sufficient oxygen and nutrient supply.

End-ischemic HMP with oxygen (HOPE) presents is marked by active oxygenation of the perfusate during MP. Even though beneficials effects of HOPE were reported in preclinical studies, no significant impact on DGF, PNF or graft survival after one year in human KT could be demonstrated. In contrast to hypothermic preservation methods, data on NMP in human KT is limited. In fact, there are no registered randomized controlled clinical trials (RCT), comparing end-ischemic NMP versus SCS in donation after brain death (DBD), the only legal donation circumstance in Germany.

The aim of this study is to investigate the impact of end-ischemic NMP compared to SCS in a multicenter prospective randomized controlled clinical trial (RCT) using ECD kidney allografts from DBD donors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients 18 years or older
* Patients suffering from end-stage kidney disease / kidney failure
* Listed for kidney transplantation
* Receiving ECD-allograft

Exclusion Criteria:

* Recipients of living donor kidney transplants
* Previous kidney transplantation
* Combined transplantations (liver-kidney, kidney-pancreas, etc.)
* Participation in other kidney related trials
* Exposure to an investigational drug within 30 days prior to inclusion
* Unwilling or unable to follow the procedures outlined in the protocol
* Mentally or legally incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Kidney function | After 6 months postoperatively
  Estimated glomerular filtration rate (eGFR)

SECONDARY OUTCOMES:
Kidney function | After 3- and 12 months postoperatively
  Estimated glomerular filtration rates (eGFR)
Delayed graft function | First 7 postoperative days
  Incidence (absolute and percentage numbers) and duration (in days) of delayed graft function (defined as the period between kidney transplant and last dialysis)
Functional delayed graft function | First 7 postoperative days
  Incidence (absolute and relative numbers) and duration (in days) of functional DGF (defined as <10% fall in serum creatinine for 3 consecutive days in the first week post-transplantation)
Creatinine change ratio | Day 2 and day 5 postoperatively
  Creatinine change ratio at day 2 (referred to day 1) and Creatinine change ratio at day 5 (referred to pretransplant serum Creatinine)
Primary non function (PNF) | After 3 months postoperatively
  Incidence of PNF descriped as persisting dialysis dependency after kidney transplantation
Incidence and severity of postoperative complications | 90-days and 1-year postoperatively
  Assessed by the Clavien-Dindo complication score and the comprehensive complication index (CCI®)
Hospitalization | Follow-up duration of 1-year
  Duration of hospital stay
Cost analysis | Follow-up duration of 1-year
  Total costs of treatment and hospital stay
Recipient- and graft survival | Follow-up duration of 1-year
  One-year recipient- and graft survival
Acute rejection incidence | Follow-up duration of 1-year
  Biopsy proven acute rejection

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Charité Universitaetsmedizin Berlin, Campus Mitte | Campus Virchow-Klinikum, Berlin
  - Medizinische Hochschule Hannover (MHH), Department of Surgery and Transplantation, Hanover
  - University Hospital Heidelberg, Department of Surgery and Transplantation, Heidelberg
  - Ludwig-Maximilian's University, Campus Grosshadern, Department of General, Visceral, and Transplant Surgery, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743
- See also: Study group webpage — http://www.hopeliver.com